CLINICAL TRIAL: NCT04338217
Title: Evaluation of the Open-bite Bionator Versus the Removable Posterior Bite Plane With a Tongue Crib in the Early Treatment of Skeletal Anterior Open Bite: A Randomized Controlled Trial
Brief Title: Early Treatment of Skeletal Anterior Open Bite by Two Appliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-02-2020
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Open Bite
MeSH Terms: conditions — Open Bite | interventions — Activator Appliances

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bionator (Experimental): The modified Bionator was used to correct the open bite malocclusion. Patients were asked to wear the appliance every day.
  Interventions: Device: Bionator
- Removable Appliance with Posterior Bite Planes (Active Comparator): A removable appliance with poster bite planes was used to correct the open bite malocclusion. Patients were asked to wear this appliance full time expect eating times.
  Interventions: Device: Removable Appliance with Posterior Bite Planes

INTERVENTIONS:
Device: Bionator — This is a functional appliance that is used to overcome the functional problems and to correct the open bite deformity
  Arms: Bionator
Device: Removable Appliance with Posterior Bite Planes — This is a one-jaw appliance that is used in conjunction with a tongue crib to control the faulty positions of the tongue and to help in closing the open bite through the use of posterior bite planes.
  Arms: Removable Appliance with Posterior Bite Planes

SUMMARY:
Open bite is a common dentoalveolar component of the facial pattern of the excessive vertical dimension patients that is also known as the gaping angle face pattern.It is a deformation in the vertical relationship between the upper and the lower dental arches that is characterized by the loss of contact between the opposite dental segments.

DETAILED DESCRIPTION:
An open bite develops as a result of the interaction of many etiologic factors, both hereditary and environmental. Prolonged sucking habits and hyper-divergent facial characteristics are significant risk factors for an anterior open bite in the mixed dentition. Abnormal tongue posture (frequently associated with enlarged adenoids or tonsils) and tongue thrust also can be involved in the establishment of alveolar and skeletal discrepancies concurrent with vertical problems Two types of an open bite are recognized in this profession: (1) dentoalveolar open bite: the abnormality formalities aspects limiting in the dental and alveolar region, usually associated with abnormal function habits as the thumb sucking and (2) Skeletal open bite: that's associated with an over high of the lower facial vertical dimension and a large plane angle of the lower jaw. open bites associated with excessive vertical skeletal dimensions are difficult to treat and tend to relapse The investigators must be recognized between the dentoalveolar open bite and the open bite caused by formalities disorders and the position disorders of the upper or the lower jaw or both. Dental an open bite can be corrected by itself if the treatment was beginning early and it's responding Easley to the mechanical treatment methods and the functional treatment approaches that depending on the muscular activity

ELIGIBILITY:
Inclusion Criteria:

* Anterior open bite (2-10) mm.
* Skeletal Class I or II malocclusion.
* MP-SN angle ranged between (33-45) degrees.
* MM angle ranged between (27-37) degrees.
* Age between 7.5-10.5 years.

Exclusion Criteria:

* Patients who had an old orthodontic treatment
* People with a syndrome or congenital deformity

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Change in the SNA angle | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This angle represents the position of upper jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken twice and this angle is going to be measured in degrees between points S, N, and A.
Change in the SNB angle | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This anglrepresents the position of lower jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken twice and this angle is going to be measured in degrees between points S, N, and B.
Change in the ANB angle | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This angle represents the spatial relationship between the upper and lower jaws in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken twice and this angle is going to be measured in degrees between A, N, and B.
Changes in the MM angle | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This angle represents the amount of vertical divergence between the upper and lower jaws in the cephalometric analysis. Lateral cephalograms will be taken twice and this angle is going to be measured in degrees between the maxillary plane and mandibular plane.
Changes in the SN-OCP angle | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This angle represents the relationship between the occlusion plane and the cranial base in the cephalometric analysis in the vertical direction. Lateral cephalograms will be taken twice and this angle is going to be measured in degrees between the SN plane (anterior cranial base plane) and the OCP (occlusal) plane.
Changes in the SN-MP angle | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This angle represents the relationship between the lower jaw plane and the cranial base in the cephalometric analysis in the vertical direction. Lateral cephalograms will be taken twice and this angle is going to be measured in degrees between the anterior cranial base plane (SN plane) and the mandibular plane (MP plane).
Changes in the SN-SPP angle | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This angle represents the relationship between the upper jaw plane and the cranial base in the cephalometric analysis in the vertical direction. Lateral cephalograms will be taken twice and this angle is going to be measured in degrees between the anterior cranial base plane (SN plane) and the maxillary plane (SPP plane).
Changes in the overbite (Ovb) | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This is a vertical measurement done on the cephalometric tracings in millimeters.
  It is the vertical overlap between the upper incisors and the lower incisors.
Changes in the overjet (Ovj) | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This is a horizontal measurement done on the cephalometric tracings in millimeters.
  It is the amount of protrusion of upper incisors in relation to the lower incisors.
Changes in the Bjork sum | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  Lateral cephalograms will be taken twice and this measurement is the sum of three different angles: (N-S-Ar + S-Ar-Go +Ar-Go-Me). These angles are well-known to orthodontists.
Changes in the N-A-Pog angle | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  Lateral cephalograms will be taken twice and this angle is going to be measured in degrees between three points: N, A, and Pogonion (Pog).
  N is located on the nasal bone. A is located at the maximum concavity of the anterior upper alveolus between the central incisors.
  Pog is the located at the most prominent point on the chin contour.
Changes in the UI- LI angle | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This angle represents the relationship between the upper and the lower incisor axes in the cephalometric analysis. Lateral cephalograms will be taken twice and this angle is going to be measured in degrees between the long axis of the upper incisor and the long axis of the lower incisor.
Changes in the NS-GN angle | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This angle represents the growth pattern of the mandible in the cephalometric analysis in the vertical direction. Lateral cephalograms will be taken twice and this angle is going to be measured in degrees between the anterior cranial base plane (NS plane) and the the Y-axis plane (i.e. the facial axis plane defined by two points: Sella Point and Gnathion 'Gn' Point).
Changes in the posterior facial height (S-Go) | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This will be vertically measured in millimeters from S point to Go point. 'S' point referes to Sella Turcica point. 'Go' point refers to the gonial angle point (located at the corner of the mandibular ramus).
Changes in the anterior facial height (N-Me) | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This will be vertically measured in millimeters from N point to Me point. 'N' point refers to the Nasion point. 'Me' point refers to the Menton point (located at the lower border of the chin).
Changes in the 'NasoLab' angle | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This angle represents the relationship between the nose and the upper lip in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken twice and this angle is going to be measured in degrees between the lower nasal tangent (i.e. the plane that touches the lower border of the columella), and the upper lip plane (i.e. the plane that goes through points Subnasale and Labrale Superius).
Changes in the 'MentoLab' angle | T1: one day before the beginning of treatment; T2: within two hours after the last treatment session
  This angle represents the relationship between the chin and the lower lip in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken twice and this angle is going to be measured in degrees between two planes: the lower lip tangent plane (from 'Labrale inferius' to mentolabial point) and upper anterior chin plane (from mentolabial point to Pogonion point).

CONTACTS AND LOCATIONS:
Overall Officials: Mahran Raheel Mousa, DDS MSc, Principal Investigator — PhD student, Orthodontics Department, University of Damascus Dental School; Hassan Farah, DDS MSc PhD, Study Chair — Professor of Orthodontics, University of Hama, Hama, Syria
Locations (1):
- Orthodontic Department, University of Al-Baath Dental School, Hama, Hamah, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torres F, Almeida RR, de Almeida MR, Almeida-Pedrin RR, Pedrin F, Henriques JF. Anterior open bite treated with a palatal crib and high-pull chin cup therapy. A prospective randomized study. Eur J Orthod. 2006 Dec;28(6):610-7. doi: 10.1093/ejo/cjl053. Epub 2006 Nov 13. PMID 17101701
- [Background] Defraia E, Marinelli A, Baroni G, Franchi L, Baccetti T. Early orthodontic treatment of skeletal open-bite malocclusion with the open-bite bionator: a cephalometric study. Am J Orthod Dentofacial Orthop. 2007 Nov;132(5):595-8. doi: 10.1016/j.ajodo.2005.12.035. PMID 18005832
- [Background] Meibodi SE, Fatahi Meybodi S, Samadi AH. The effect of posterior bite-plane on dentoskeletal changes in skeletal open-bite malocclusion. J Indian Soc Pedod Prev Dent. 2009 Oct-Dec;27(4):202-4. doi: 10.4103/0970-4388.57653. PMID 19915269
- [Background] Cozza P, Baccetti T, Franchi L, Mucedero M. Comparison of 2 early treatment protocols for open-bite malocclusions. Am J Orthod Dentofacial Orthop. 2007 Dec;132(6):743-7. doi: 10.1016/j.ajodo.2005.11.045. PMID 18068591
- [Background] Mucedero M, Vitale M, Franchi L, Cozza P, Perillo L. Comparisons of two protocols for early treatment of anterior open bite. Eur J Orthod. 2017 Jun 1;39(3):270-276. doi: 10.1093/ejo/cjw039. PMID 27141934
- [Background] Cozza P, Baccetti T, Franchi L, McNamara JA Jr. Treatment effects of a modified quad-helix in patients with dentoskeletal open bites. Am J Orthod Dentofacial Orthop. 2006 Jun;129(6):734-9. doi: 10.1016/j.ajodo.2006.02.004. PMID 16769491
- [Background] Rossato PH, Fernandes TMF, Urnau FDA, de Castro AC, Conti F, de Almeida RR, Oltramari-Navarro PVP. Dentoalveolar effects produced by different appliances on early treatment of anterior open bite: A randomized clinical trial. Angle Orthod. 2018 Nov;88(6):684-691. doi: 10.2319/101317-691.1. Epub 2018 Jun 18. PMID 29911909
- [Background] Giuntini V, Franchi L, Baccetti T, Mucedero M, Cozza P. Dentoskeletal changes associated with fixed and removable appliances with a crib in open-bite patients in the mixed dentition. Am J Orthod Dentofacial Orthop. 2008 Jan;133(1):77-80. doi: 10.1016/j.ajodo.2007.07.012. PMID 18174075
- [Derived] Mousa MR, Hajeer MY, Farah H. Evaluation of the open-bite Bionator versus the removable posterior bite plane with a tongue crib in the early treatment of skeletal anterior open bite: A randomized controlled trial. J World Fed Orthod. 2021 Dec;10(4):163-171. doi: 10.1016/j.ejwf.2021.08.001. Epub 2021 Aug 27. PMID 34462242